CLINICAL TRIAL: NCT04122612
Title: Prenatal and Postnatal Determinants in Shaping Offspring's Microbiota in the First Year of Life: A Study Protocol
Brief Title: Shaping Microbiome in the First 1,000 Days of Life
Acronym: AMAMI
Status: Completed | Type: Observational
Sponsor: University of Pavia (Other)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other); Istituti Clinici Scientifici Maugeri SpA (Other); Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Responsible Party: Principal Investigator, Hellas Cena, Professor, University of Pavia
Other Study IDs: 20191004
Record Dates: First submitted 2019-10-07; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Microbial Colonization
Keywords: microbiota; 1000 days; maternal lifestyle; diet; pregnancy
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fecal and urine sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Events occurring in the early stages of life play an important role in the development of chronic diseases; diet and lifestyle during pregnancy are recognized to be crucial determinants in modulating offspring microbiota, throughout a vertical transfer of dysbiotic maternal ambient. Moreover, the intestinal colonization is maximized in the first two years of life through newborn's type and time of feeding. This study will provide the starting point for a future prospective observational study to assessing the association between maternal lifestyle with infant microbiota and their influence future health.

DETAILED DESCRIPTION:
Evidence from the Developmental Origins of Health and Disease (DOHaD) theory has pointed out biological mechanisms supporting the intergenerational nature of non communicable diseases (NCDs), which are an increasing public health problem in many countries. Furthermore, scientific evidence confirms that the events occurring in the early stages of life play a critical role in fostering the development of chronic diseases (e.g. overweight and obesity, allergies, cardiovascular and metabolic diseases, neurocognitive impairment and cancers), throughout the life-course, indicating the high relevance of "the maternal environment" impact on the life of the future child. This crucial window goes from the conception to the two years of life, and it is known as 'first thousand days'.

Nutritional status during pregnancy is one of the crucial determinants in modulating the characteristics of the "maternal environment" in which the foetus originates and develops. Therefore, adequate nutrition just before conception, during pregnancy, infancy and early childhood is essential to ensure growth, health, and development of children to their full potential.

Epigenetic links have been confirmed in mice between the prenatal diet and the increased incidence of obesity, type 2 diabetes and other metabolic associated conditions in their offspring. However, specific epigenetic regulation mechanisms are still unclear. Recently, an increasing number of animal and human studies have proposed the hypothesis that the gut microbiota may be considered an important mediator of vital microbiome-host interaction(s) under health or disease conditions. Moreover, microbiota has been shown to pass features from one generation to the next via maternal contact; in fact, recent observation of microbial presence in placenta, meconium and amniotic fluid has suggested a significant interplay between the environmental microbes and the developing gastrointestinal tract of the fetus even before delivery. Thus, the alteration of microbiota composition, driving to increased long-term susceptibility to diseases, can begin early in life.

Examination of the neonatal gut microbiome immediately after delivery revealed that it varied by virtue of maternal gestational diet suggesting that the colonization of the infant gut is likely to occur prior to parturition.

During the first months after birth, the bacterial flora in the gut is known to be affected by many factors, including mode of delivery, use of antibiotics or probiotics, geographical location, type and time of feeding.

Moreover, maternal exposures during pregnancy to several environmental chemicals are known to induce perturbations in the composition of the gastrointestinal microbiome. Among these substances, endocrine disruptor chemicals (EDCs), such as phthalates, bisphenol and hydroxypyrene, which can be found in oil and water resistant textile coatings, non-stick cookware, food container coatings, floor polish, fire-fighting foam, and industrial surfactants, are a class of suspected obesogenic contaminants persisting in the environment and humans. EDCs have been also detected in cord blood samples, suggesting that exposure starts prenatally and early life EDC exposures may perturb neuroendocrine systems involved in growth, energy metabolism, appetite, adipogenesis, and glucose-insulin homeostasis promoting childhood obesity development.

After this first period, the gut microbial composition continues to evolve until the age of 2-3 years; these first years represent as "a window of opportunity" for microbial modulation, influenced by complementary feeding period, gradual transition from milk-based infant feeding to weaning and solid foods, usually occurring between 6 and 24 months.

A.MA.MI is a longitudinal, prospective, observational study that includes a group of mother-infant pairs (n=60) attending the Neonatal Unit, Fondazione IRCCS Policlinico San Matteo, Pavia (Italy). The study was planned to provide data collected before discharge (T0) and at 1,6,12 months after birth (T1,T2,T3). Maternal and infant anthropometric measurements are assessed at each time. Other variables evaluated are pre-pregnancy/gestational weight status (T0), maternal dietary habits/physical activity (T1-T3); infant medical history, type of feeding, antibiotics/probiotics/supplements use, environment exposures (e.g cigarette smoking, pets, environmental temperature) (T1-T3). A child stool sample was planned to be collected at each time and analyzed using metagenomics 16S ribosomal RNA gene sequence-based methods. Maternal urine samples were planned to be collected at T3 to investigate pollutants exposure (Phthalates, Bisphenol A and Hydroxypyrene).

Since there are still limited knowledge about the child's microbiota, its changes over time and the host and environmental interactions in shaping its composition, further prospective studies are needed to determine how different factors related to diet-related factors, lifestyle, drugs and anthropometric measures can influence microbial colonization of the gut during early childhood and influence the future health status.

ELIGIBILITY:
Inclusion Criteria:

* Infants of both sexes born to natural or caesarean delivery;
* Gestational age between 35 and 42 completed weeks;
* Italian-speaking parents;
* Ability of the parent/guardian to give informed consent;
* Ability of the mother to respond to the structured interview/questionnaires;

Exclusion Criteria:

Children or mothers with genetic/congenital diseases;

* Children hospitalized immediately after birth;
* Children selected for other clinical studies;
* Presence of gestational diabetes;
* Presence of hyperthyroidism during pregnancy;
* Parents refusing to sign the informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 60 dyads (mother/new-born) attending the Neonatal Unit, Fondazione IRCCS Policlinico San Matteo, Pavia (Italy)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-09-23 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Change in intestinal microbiota composition from 0 to 12 months of life | 0 months (2-3 days after birth); 1 months after birth; 6 months after birth; 12 months after birth.
  Investigate the intestinal microbiota development of infants at 0, 1, 6, 12 months after birth by:
  i) Identifying the relative abundance of the dominant organism genera; ii) Assessing the microbial diversity (α-diversity); iii) Assessing inter-individual variation (β-diversity).

SECONDARY OUTCOMES:
examine the association of maternal and infants factor and the intestinal microbiota development of infants. | 0 months (2-3 days after birth); 1 months after birth; 6 months after birth; 12 months after birth.
  exploring the possible correlation between maternal factors before pregnancy (weight status), gestational exposures (maternal diet, physical activity, weight status, EDCs), mode of delivery, lactation (formula or breastfeeding), family environment exposure, infant diet, sleeping habits and infant intestinal microbiota composition, during the first year of life at different follow-up:
  * immediately after the delivery (not more than 2-3 days after the delivery, T0);
  * 1 month after birth (T1);
  * 6 months after birth (T2);
  * 12 months after birth (T3).

CONTACTS AND LOCATIONS:
Overall Officials: Hellas Cena, Principal Investigator — Università di Pavia
Locations (1):
- IRCCSSMP, Pavia, Italy

REFERENCES:
- [Derived] Vacca M, Raspini B, Calabrese FM, Porri D, De Giuseppe R, Chieppa M, Liso M, Cerbo RM, Civardi E, Garofoli F, Cena H, De Angelis M. The establishment of the gut microbiota in 1-year-aged infants: from birth to family food. Eur J Nutr. 2022 Aug;61(5):2517-2530. doi: 10.1007/s00394-022-02822-1. Epub 2022 Feb 25. PMID 35211851
- [Derived] Raspini B, Porri D, De Giuseppe R, Chieppa M, Liso M, Cerbo RM, Civardi E, Garofoli F, Monti MC, Vacca M, De Angelis M, Cena H. Prenatal and postnatal determinants in shaping offspring's microbiome in the first 1000 days: study protocol and preliminary results at one month of life. Ital J Pediatr. 2020 Apr 15;46(1):45. doi: 10.1186/s13052-020-0794-8. PMID 32293504